CLINICAL TRIAL: NCT00490386
Title: Alkoholihaimatulehduksen Uusiminen
Brief Title: Helicobacter Pylori and Acute Alcohol Induced Pancreatitis
Status: Completed | Type: Observational
Sponsor: Tampere University (Other)
Other Study IDs: R00126-1
Record Dates: First submitted 2007-06-20; First posted 2007-06-22 (Estimated); Last update posted 2007-06-22 (Estimated); Status verified 2007-06

CONDITIONS: Pancreatitis, Acute; Helicobacter Infections
Keywords: Retrospective; Length of Stay; Helicobacter pylori
MeSH Terms: conditions — Pancreatitis; Helicobacter Infections

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Other
Oversight: Data Monitoring Committee: No

SUMMARY:
This study is performed to measure wether Helicobacter Pylori has an effect on the incidence and course of acute alcohol induced pancreatitis

DETAILED DESCRIPTION:
A recent pilot study unexpectedly discovered, that Helicobacter pylori infection was rare in patients having their first acute alcohol induced pancreatitis (AAIP) when compared to subjects with similar alcohol use but no history of pancreatitis. This subject has not been studied in humans until now. Therefore we seek to study, with a larger material, wether AAIP is associated with lower prevalence of Helicobacter pylori, by measuring the antibodies against Helicobacter pylori from the sera of AAIP patients and from a control group of alcoholics with no history of AAIP.

ELIGIBILITY:
Inclusion Criteria:

* Acute alcohol pancreatitis (first)

Exclusion Criteria:

* Death during hospitalization

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2006-06

CONTACTS AND LOCATIONS:
Overall Officials: Jahangir A Khan, MS, Principal Investigator — Department of Gastroenterology and Alimentary Tract Surgery, Tampere University; Isto Nordback, MD, Study Director — 1Department of Gastroenterology and Alimentary Tract Surgery, Tampere University Hospital
Locations (1):
- Tampere University Hospital, Tampere, Pirkanmaa, Finland

REFERENCES:
- [Background] Pelli H, Herzig KH, Uotila S, Raty S, Laine S, Sand J, Nordback I. Duodenal diazepam-binding protein expression and plasma cholecystokinin after alcoholic pancreatitis. Scand J Clin Lab Invest. 2006;66(8):677-83. doi: 10.1080/00365510600930918. PMID 17101560